CLINICAL TRIAL: NCT06812325
Title: A Randomized, Double-masked, Controlled, Safety and Tolerability Study of VRDN-003 in Participants With Thyroid Eye Disease (TED)
Brief Title: A Safety and Tolerability Study of VRDN-003 in Participants With Thyroid Eye Disease (TED)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRDN-003-303
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Eye Disease (TED)
Keywords: Graves; Thyroid Eye Disease; Thyroid-Associated Ophthalmopathy; Dysthyroid Ophthalmopathy; Graves Eye Disease; Graves Orbitopathy; Myopathic Ophthalmopathy; Congestive Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the two study arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Site personnel (except pharmacy personnel preparing the injection), and Sponsor are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VRDN-003 every 4 weeks (Experimental): 6 subcutaneous administrations of VRDN-003
  Interventions: Drug: VRDN-003
- VRDN-003 every 8 weeks (Experimental): 3 subcutaneous administrations of VRDN-003 and 3 subcutaneous administrations of placebo
  Interventions: Drug: VRDN-003; Drug: Placebo

INTERVENTIONS:
Drug: VRDN-003 — VRDN-003 is an investigational, subcutaneously administered, humanized monoclonal antibody directed against the Insulin-like Growth Factor-1 receptor (IGF-1R).
Drug: Placebo — Placebo injections that appear identical to VRDN-003 injections but have no active drug.
  Arms: VRDN-003 every 8 weeks

SUMMARY:
This is a clinical trial assessing the safety and tolerability of an investigational drug, VRDN-003, in participants with Thyroid Eye Disease (TED).

DETAILED DESCRIPTION:
This is a randomized (meaning participants will be assigned to study arms by chance), double-masked (meaning study doctor and participant will not know which study arm participant is assigned to), controlled study that will include participants with TED of any duration. The key objectives of this study are to determine if VRDN-003 is safe and tolerable when administered as a series of subcutaneous (SC) injections every 4 weeks or every 8 weeks in participants with TED.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a clinical diagnosis of TED with or without proptosis and with any CAS (0-7) and in the opinion of the Investigator may benefit from VRDN-003
* Not require immediate ophthalmological or orbital surgery in the study eye for any reason.
* Must agree to use highly effective contraception as specified in the protocol
* Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria:

* Must not have received prior treatment with another anti-IGF-1R therapy
* Must not have received systemic corticosteroids or steroid eye drops for any condition, including TED, or selenium within 2 weeks prior to first dose.
* Must not have received other immunosuppressive drugs for any condition, including TED, or any other therapy for TED within 12 weeks prior to first dose
* Must not have received an investigational agent for any condition, including TED, within 8 weeks or longer duration (depending on the type of investigational agent) prior to first dose
* Must not have received radioactive iodine (RAI) treatment within 8 weeks prior to first dose
* Must not have had previous orbital irradiation or decompression surgery for TED to the study eye's orbit
* Must not have a pre-existing ophthalmic condition in the study eye which in the study doctor's opinion, would interfere with interpretation of study results
* Must not have abnormal hearing test before first dose. Must also not have a history of ear conditions considered significant by study doctor
* Must not have a history of inflammatory bowel disease
* Female TED participants must not be pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event (TEAE) incidence rate through Week 24 | Week 24
  Treatment Emergent Adverse Event (TEAE) incidence rate through Week 24

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye at Week 24 as measured by exophthalmometer | Week 24
  Change from baseline in proptosis in the study eye
TEAE incidence rate through Week 52 | Week 52
  Treatment Emergent Adverse Event (TEAE) incidence rate measurement through Week 52

CONTACTS AND LOCATIONS:
Locations (64):
- United States (32):
  - Catalina Eye Care, Tuscon, Arizona
  - United Medical Research Institute, Inglewood, California
  - Orbital Plastics, Newport Beach, California
  - California Eye Specialists Medical Group INC, Pasadena, California
  - FOMAT Medical Research, Pismo Beach, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - Pacific Neuroscience Institute at Saint John's Physician Partners, Torrance, California
  - C A Clinical Trial Corp., Cape Coral, Florida
  - Herco Medical and Research Center, Coral Gables, Florida
  - Alfa Medical Research, Davie, Florida
  - D H Doral Research Center, Doral, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - Sina Medical Center, Homestead, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Southern Clinical Research LLC, Miami, Florida
  - Retreat Medical Research, Miami, Florida
  - Continental Clinical Research, Miami, Florida
  - Edward Jenner Research Group LLC, Plantation, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Advanced Quality Medical Research, Orland Park, Illinois
  - Ophthalmic Consultants of Boston, East Weymouth, Massachusetts
  - Fraser Eye Care Center, Fraser, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Missouri Kansas City, Kansas City, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Jackson Clinic, Jackson, Tennessee
  - DFW Clinical Trials, Carrollton, Texas
  - Neuro Eye Clinical Trials, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - Eyeplastx, San Antonio, Texas
  - Elevate Clinical Research, Seabrook, Texas
- France (3):
  - Servicde d'Endocrinologie, Diabetologieet Nutrition Centre Hospitalier Universitaire d'Angers, Angers
  - Abeillon du Payrat, Bron
  - Hôpital La Pitiélsalpêtrière, Paris
- Germany (4):
  - Charite Universitatsmeizin Berlin KoR Campus Virchow Klinikum, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitaetsmedizin Goettingen, Göttingen
  - Johannes Gutenberg University Medical Center Department of Medicine 1, Mainz
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Klinika Okulistyki, Centrum Badań Klinicznych, Bialystok
  - Optimum Profesorskie Centrum Okulistyki Sp. z o. o., Gdansk
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Santa Familia PTG Lodz, Lodz
  - ETG Lublin, Lublin
  - Centrum Medyczne Pulawska Sp. z o.o., Piaseczno
  - Warszawski Szpital Okulistyczny, Warsaw
  - Polimedica PTG, Warsaw
- Spain (7):
  - Hospital Provincial de Conxo, A Coruña
  - Institut Català de Retina, Barcelona
  - Hospital La Arruzafa, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarre, Navarrés
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet Consultas de Oftalmologia, Zaragoza
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty Hospital, Ankara
  - Hacettepe Univeristy Medical Fculty Hospital, Ankara
  - Akdeniz Üniversitesi Tıp Fakültesi Göz Hastalıkları Anabilim Dalı, Antalya
  - Marmara Üniversitesi Pendik Eğitim ve Araştırma Hastanesi Göz Hastalıkları Kliniği, Istanbul
- United Kingdom (6):
  - University Hospitals Bristol and Weston NHS Foundation Trust Clinical Research Unit, Bristol
  - Addenbrookes Hospital, Cambridge
  - Imperial College Healthcare NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Moorefields Eye Hospital NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle